CLINICAL TRIAL: NCT01891630
Title: Observational Assessment of Baseline Asthma Control as a Susceptibility Factor for Air Pollution Health Effects in African-American Children With Moderate-severe Asthma (Teen AIRE Study)
Brief Title: Observational Assessment of Baseline Asthma Control in African-American Children
Acronym: TeenAire
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michelle Hernandez, MD, Dr. Hernandez, University of North Carolina, Chapel Hill
Other Study IDs: 12-1588
Record Dates: First submitted 2013-06-25; First posted 2013-07-03 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Asthma
Keywords: African American; Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AA children: African-American children with moderate-to-severe asthma living in a defined geographical area whose asthma is poorly controlled, and up to 30 moderate-to-severe African-American asthmatic children living in the same defined geographical area whose asthma is well controlled.

SUMMARY:
To determine if baseline asthma control influences susceptibility to pollutant-induced health effects in African-American children with moderate-to-severe asthma.

DETAILED DESCRIPTION:
In the general public, certain sub-populations are at higher risk for adverse health effects due to air pollution exposure. Asthmatics have been identified as one such susceptible population due to the observed association of elevated air pollution levels and increased incidences of acute asthma exacerbations as evidenced by decreased lung function values and respiratory symptoms, shortness of breath, emergency department (ED) visits, and hospitalizations (6-13). A study conducted by Mar et al (2004) reported that health outcomes associated with coarse particulate matter (PM2.5-10) were more notable in children with asthma than in adults with asthma (14) and a large epidemiological study of asthmatic children in the Northeastern US showed that asthma morbidity on high ozone days was consistently highest among children age 6 to 18 years (15). Furthermore, children with persistent asthma (requiring daily maintenance medication) were shown to be at increased risk of respiratory symptoms and rescue medication use after ambient ozone exposure compared to children with mild intermittent asthma (16). Together, these studies demonstrate an additional level of susceptibility to air pollution in children compared with adults and in children with persistent asthma compared with mild intermittent asthma.

African-American patients appear to be particularly susceptible to asthma-related complications, with rates of asthma-related emergency department visits, hospitalizations, and death approximately 2 to 3 times the rates found in Caucasian subjects (17) . Furthermore, a higher proportion of African-American asthmatics have poorly-controlled asthma compared to non-African-American asthmatics (18). In a recent pediatric study, very poorly controlled asthmatics had an increased risk of asthma-related hospitalization, emergency department visits, or corticosteroid burst (OR, 6.4; 95% CI, 1.2-34.5) compared with those whose asthma was under better control over a 2-year period (19).

The goal of this panel study is to determine if African-American children with poorly-controlled moderate-to-severe persistent asthma are at increased risk for cardiopulmonary effects as a result of ambient air pollution exposure compared to age- and race-matched well-controlled moderate-to-severe asthmatic children. The primary cohort for this panel study will be African-American children between the ages of 12-17 years with moderate-to-severe asthma (divided between the study populations of poorly-controlled asthma and well-controlled asthma). Since this study is exclusively focused on an African-American population, it is not designed to address the effect of race/ethnicity on baseline asthma control. Volunteers will be recruited primarily from the UNC Pediatric Pulmonary clinic and the UNC Allergy/Immunology clinic located at Rex Hospital in Raleigh, NC in which Dr. Hernandez is an attending physician. These volunteers are well-characterized asthmatics followed regularly by a pediatric pulmonologist (Dr. Ceila Loughlin) and by a pediatric allergist (Dr. Michelle Hernandez) at the Rex location. In order to ensure that the two cohorts experience equivalent daily exposures to ambient air pollutants, the study population will be recruited from a defined geographical region within a reasonable driving distance of the Rex Hospital and in relative proximity to the state-operated monitoring station for ambient air pollutants.

Establishing a relationship between asthma control and adverse health outcomes in response to air pollution exposure will provide health care providers and parents of children with moderate-to-severe asthma the information necessary to take proactive action on high air pollution days as they are communicated to the public through color-coded days based on the National Ambient Air Quality Standards (NAAQS) established by the EPA. If asthma control is determined in this study to be a risk factor for susceptibility, future work will be directed toward establishing the mechanism underlying the susceptibility which may then lead to the potential design of new therapies or intervention strategies.

ELIGIBILITY:
Inclusion Criteria for all subjects:

1. Self-identified as African-American
2. Ages 12-17 years
3. Live within convenient driving distance of the UNC Rex Clinic in Raleigh, NC.
4. Physician-diagnosis of moderate-to-severe persistent asthma
5. Current treatment with appropriate therapy for moderate-to-severe persistent asthma symptoms as per the NHLBI guidelines including: Daily controller medication use for asthma requiring at least a medium-dose inhaled corticosteroids (ICS) or a low dose ICS + long-acting beta2 agonist (LABA) combination. Subjects may use daily or every other day oral corticosteroids for control of asthma symptoms

Inclusion criteria for well-controlled asthmatics (from NHLBI guidelines):

1. Nighttime awakening with asthma symptoms ≤ 2x/month over the past 6 months
2. Use of short-acting beta2 agonist for symptom control ≤ 2 days /week over the past 6 months
3. Asthma Control Test score >19. The Asthma Control Test is a standardized clinical tool to assess asthma control over the previous 4 week period (attached).
4. Baseline FEV1(pre-albuterol) > 80% of that predicted for gender, ethnicity, age and height (NHANES III predicted set)

Inclusion criteria for poorly-controlled asthmatics (from NHLBI guidelines):

1. Nighttime awakening with asthma symptoms > 2x/month over the past 6 months
2. Use of short-acting beta2 agonist for symptom control > 2 days /week over the past 6 months
3. Asthma Control Test score <19. The Asthma Control Test is a standardized clinical tool to assess asthma control over the previous 4 week period (attached).
4. Baseline FEV1 (pre-albuterol) < 80% of that predicted for gender, ethnicity, age and height (NHANES III predicted set)

Exclusion criteria for all subjects:

1. Children younger than age 12 and older than 17
2. Children unable to perform spirometry
3. Medical history or underlying health problems that may preclude participation in the protocol per the study physician (including but not limited to cystic fibrosis, chronic bronchitis, recurrent pneumonia, immunodeficiency, hematologic disorders)
4. History of bleeding disorder or anemia
5. Subjects and families unwilling to travel to the clinic for the required 6 visits
6. Unwilling or unable to refrain from the following medications for the week prior to the study as well as the week of the study including fish oil; anti-inflammatory agents such as ibuprofen (Advil, Motrin), naproxen (Aleve) or aspirin as needed**. Acetaminophen (Tylenol) is allowed.**If the child requires anti-inflammatory medications for a fever or joint/muscle pain, in the week prior to the study visit, all subsequent visits may be rescheduled.
7. Other uncontrolled health problems
8. Non-English speaking subjects

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We will enroll a maximum of 60 African-American children with moderate-to-severe persistent asthma in which half of the cohort will have well-controlled asthma and the other half will have poorly-controlled asthma (defined by NHLBI guidelines). Participants will be of both genders, ages 12-17 years old, and live within a convenient driving distance from the study site located within the UNC Pediatric Pulmonary and UNC Pediatric Allergy and Immunology Subspecialty clinics at Rex Hospital located in Raleigh, NC.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in lung function assessed by spirometry over a period of 6-8 weeks | at each weekly study visit over 6-8 weeks
  FEV1, FVC and FEV1/FVC ratio

SECONDARY OUTCOMES:
Asthma Control Composite Measure | at each weekly study visit over 6-8 weeks
  The following measures will be used to assess overall asthma control:
  1. . asthma control questionnaire score.
  2. . Number of urgent care visits for asthma during the interval study period.
  3. . requirement for oral steroid use for asthma during the interval study period.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hernandez, MD, Principal Investigator — UNC
Locations (1):
- Rex Hospital, Raleigh, North Carolina, United States